CLINICAL TRIAL: NCT06570044
Title: Evaluation of PerioMonitor for Detection of Oral Inflammatory (OI) in Human Subjects in Medical Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oral Science International Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20240513
Record Dates: First submitted 2024-08-19; First posted 2024-08-26 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Oral Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- PerioMonitor (Experimental)
  Interventions: Diagnostic Test: PerioMonitor

INTERVENTIONS:
Diagnostic Test: PerioMonitor — Collection of oral rinse specimen and perform the PerioMonitor test as per the method described in the instructions for use

SUMMARY:
The purpose of the study is to evaluate the usability of PerioMonitor™ in a medical clinic environment and to evaluate the effectiveness of a referral system from physicians to dentists for patients identified with high oral inflammation.

PerioMonitor™ is an In Vitro Diagnostic (IVD) device intended as an aid in the detection of oral inflammation in individuals of 18 years and older. This test is intended for use at point-of-care (POC) sites by health care professionals (e.g., physicians, nurses, medical assistants, dentists, dental hygienists, and dental assistants).

ELIGIBILITY:
Inclusion Criteria:

* subject fluent in English
* subject has signed the ICF

Exclusion Criteria:

* subject with altered mental status/inability to provide informed consent or follow the procedure of the Study
* Previous enrolment into the current Study
* Patients with known severe oral diseases such as oral cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Ratio (%) of valid tests/performed tests | Day 0
  The ratio of valid PerioMonitor tests (with no issue reported) over the total number of tests performed
Ease of Test Performance | Day 0
  The Ease-of-Test Performance will be evaluated by a 5-question questionnaire
Use error | Day 0
  Any issue encountered with collection of specimens and/or test reading. The overall ratio (%) of tests with use errors as well as the ratio per operator will be measured
Comfort to participants | Day 0
  Comfort to participants with sample collection (Yes/No). The Overall ratio (%) of discomfort ('No') as well as the ratio per operator will be measured.

SECONDARY OUTCOMES:
Proportion (%) of participants referred to a Dental Specialist | 6-Month
  The recommended course of action further to completion of the PerioMonitor test will be documented with a 4-item report form. The ratio (%) of participants referred to a dental specialist visit as the recommended course of action will be calculated.
Proportion (%) participants referred to a Dental Specialist | 12-Month
  The recommended course of action further to completion of the PerioMonitor test will be documented with a 4-item report form. The ratio (%) of participants referred to a dental specialist visit as the recommended course of action will be calculated.
Proportion (%) of compliant participants with the recommended visit to a Dental Specialist | 6-Month
  Visits to a Dental Specialist will be monitored by querying participants' electronic medical records or by direct contact (email or phone) and data (visit date, treatment) will be documented in a report form.
  The ratio (%) of participants who completed a visit to a Dental Specialist over all participants referred to a dental specialist visit as the recommended course of action will be calculated.
Proportion (%) of compliant participants with the recommended visit to a Dental Specialist | 12-Month
  Visits to a Dental Specialist will be monitored by querying participants' electronic medical records or by direct contact (email or phone) and data (visit date, treatment) will be documented in a report form.
  The ratio (%) of participants who completed a visit to a Dental Specialist over all participants referred to a dental specialist visit as the recommended course of action will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel B Low, Principal Investigator — University of Florida
Locations (1):
- 1st Family Medicine, Buckeye, Arizona, United States

IPD SHARING:
Plan to Share IPD: No